CLINICAL TRIAL: NCT01786395
Title: Phase III Clinical Study of UF-021 for Retinitis Pigmentosa - Evaluation for a Comparative Double Masked Placebo Controlled Study Period and a Continuous Administration Period
Brief Title: Phase III Efficacy and Safety Clinical Study of UF-021 for Treatment of Retinitis Pigmentosa
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: R-Tech Ueno, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UF-021-C003
Record Dates: First submitted 2013-01-23; First posted 2013-02-08 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2013-03

CONDITIONS: Retinitis Pigmentosa
Keywords: UF-021; unoprostone; rp
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — isopropyl unoprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- - UF-021 (Experimental): UF-021 is experimental code for isopropyl unoprostone
  Interventions: Drug: UF-021
- - Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UF-021
  Other Names: isopropyl unoprostone (JAN)
  Arms: - UF-021
Drug: Placebo
  Arms: - Placebo

SUMMARY:
This study is a multicenter trial performed in Japan, consisting of a comparative study period and a continuous administration period.

Effect of 0.15% UF-021 eye drops on improvement in central retinal sensitivity with HFA will be verified in 52 weeks comparative study period by a placebo-controlled, double-masked study in patients with retinitis pigmentosa.

The safety of same eye drops will also be examined in 52 weeks continuous administration period, in all the patients who completed the comparative study period.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20 years or more, 70 years or less (at obtaining informed consent)
2. Medical examination classification: Outpatients
3. Observation, examination, and surveillance in accordance with the study protocol are judged to be feasible.
4. ETDRS visual acuity test is judged to be feasible at a distance of 4 meters.
5. HFA (10-2) test is judged to be feasible by investigator.
6. Goldmann perimetry shows concentric central visual field loss (including a ring scotoma) with the central 30 degrees or less.
7. The difference in the mean retinal sensitivity at four central points must be less than 3 dB between two reliable measurements with HFA (10-2) (SITA-Standard) conducted within 31 days and both values are worse than 30 dB.(When this criterion is not met after two tests, a 3rd measurement will be implemented within 31 days from the 2nd test. The difference between the 3rd reliable measurement value and the 1st or 2nd measurements must be less than 3 dB, and both values are worse than 30 dB; the most recent data will be regarded as the data acquired before instillation.)

Exclusion Criteria:

1. Judged to have difficulty by investigator for visiting the hospital and returning home safely over the study period.
2. Planning to undergo an ophthalmic operation for eye for efficacy evaluation during study period.
3. Current treatment for glaucoma or ocular hypertension.
4. Prior ophthalmectomy or evisceration of an eye
5. Intraocular surgery within the past five months.
6. History of allergy to drugs (instillation narcotics, fluorescein, etc.) that will be used during the clinical study, and to drugs similar to the investigational product
7. Complications of diabetic retinopathy.
8. Complications of external eye inflammation, infectious diseases, or severe dry eye.
9. Use of isopropyl unoprostone in the past or present.
10. Use of the following drugs within 31 days before obtaining informed consent. Calcium antagonists, Dark adaptation improvement drug (helenien)
11. Participation in UF-021 phase Ⅱ trial (including subjects assigned to the placebo group).
12. Participation in other clinical studies within the past 6 months (However, any subject who has not been administered an investigational product will be accepted)
13. Pregnancy or the possibility of becoming pregnant. Currently breastfeeding. Childbearing patients who wish to become pregnant during the clinical study period and are not using appropriate contraceptive measures.
14. Cone-rod dystrophy where cone function was primarily impaired
15. History of optic nerve disease in the eye for efficacy evaluation
16. Complications of a moderate or more severe (grade 3 of the Emery classification) central cataract, an anterior subcapsular cataract, a posterior subcapsular cataract, and posterior capsule opacification that may exert a major influence on visual acuity in the eye for efficacy evaluation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2013-03; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Changes in the value of the mean retinal sensitivity at four central points through HFA (10-2) | baseline and 1 year

SECONDARY OUTCOMES:
- Changes in the value of the retinal sensitivity through HFA (10-2) (MD value, mean retinal sensitivity at 12 central points /24 central points /68 central points) | baseline and 1 year
- Changes in the value of the ETDRS visual acuity | baseline and 1 year
- Changes in the VFQ-25 (composite 8) value | baseline and 1 year
- Changes in the Goldmann visual field area within V4e isopter | baseline and 1 year
- Changes in the value of retinal thickness through OCT | baseline and 1 year

CONTACTS AND LOCATIONS:
Locations (34):
- Japan (34):
  - Nagoya, Aichi-ken
  - Hirosaki, Aomori
  - Chiba, Chiba
  - Matsuyama, Ehime
  - Fukuoka, Fukuoka
  - Maebashi, Gunma
  - Kure, Hiroshima
  - Sapporo, Hokkaido
  - Kobe, Hyōgo
  - Mito, Ibaraki
  - Morioka, Iwate
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Tsu, Mie-ken
  - Sendai, Miyagi
  - Miyakonojō, Miyazaki
  - Miyazaki, Miyazaki
  - Beppu, Oita Prefecture
  - Okayama, Okayama-ken
  - Tamano, Okayama-ken
  - Osaka, Osaka
  - Sayama, Osaka
  - Izumo, Shimane
  - Hamamatsu, Shizuoka
  - Ohtawara, Tochigi
  - Tokushima, Tokushima
  - Bunkyo-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Itabashi-ku, Tokyo
  - Minato-ku, Tokyo
  - Mitaka, Tokyo
  - Toyama, Toyama
  - Wakayama, Wakayama
  - Chūō, Yamanashi